CLINICAL TRIAL: NCT00580476
Title: Assessing Depression in a Geriatric Cancer Population
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: City of Hope National Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-100
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 150 patients will be women with breast cancer (75 early stage and 75 late stage)
- 2: 150 will be men with prostate cancer (75 early stage and 75 late stage)

SUMMARY:
The goal of this study is to learn more about how we measure depression in elderly cancer patients (patients aged 70 and older). Depression is one of the most common causes of emotional distress in the elderly and continues to be under-recognized. This is a problem because depression can have a negative impact on quality of life. The symptoms of depression are linked to poor health outcomes and higher costs of health care. In fact, depression is one of the top five concerns facing the elderly today.

DETAILED DESCRIPTION:
We have a few questionnaires that have been used to measure depression, but we do not know how these measures work with people with cancer. This study will help us answer this question. To complete this study, we need people who may or may not be feeling down or depressed.

If you choose to take part, you will be asked to do the following:

1. Fill out questionnaires that ask about:

   * Your age, eduction, race, and income
   * Your mood

   In all, these questionnaires will take about 10 minutes to complete.
2. Answer questions about your mood. This will also take about 10 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Age 70 and older
2. Diagnosis of early or late stage prostate cancer, or diagnosis of early or late stage breast cancer
3. Actively engaged in one of the following cancer treatments: chemotherapy, radiation therapy, hormone therapy
4. Able to provide informed consent
5. Ability to converse, write and read English

Exclusion Criteria:

1.Major psychopathology or cognitive impairment likely in the judgment of the research staff to interfere with the participation or completion of the protocol.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric Patients with Breast or Prostate Cancer
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2006-09-12 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Test the sensitivity and specificity of the Geriatric Depression Scale-Short Form and two other widely used assessments of depression to detect major and minor depression in a geriatric breast and prostate cancer population. | 2 years

SECONDARY OUTCOMES:
To develop a cut-off score for the GDS that is specific to a cancer population. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, Ph.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org